CLINICAL TRIAL: NCT06039189
Title: A Phase 3b, Multicenter, Randomized, Double-blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Guselkumab Versus Placebo for the Treatment of Low Body Surface Area (BSA) Moderate Plaque Psoriasis With Special Site Involvement
Brief Title: Study of Guselkumab Versus Placebo for the Treatment of Low Body Surface Area Moderate Plaque Psoriasis
Acronym: SPECTREM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109328; CNTO1959PSO3017 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Moderate Plaque Psoriasis
MeSH Terms: interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Guselkumab (Experimental): Participants will receive guselkumab by subcutaneous injection with placebo as needed to maintain the blind.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 2: Placebo (Placebo Comparator): Participants will receive placebo by subcutaneous injection then receive guselkumab by subcutaneous injection.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered as subcutaneous injection.
  Other Names: CNTO1959; Tremfya
Drug: Placebo — Placebo will be administered as subcutaneous injection.

SUMMARY:
The purpose of this study is to evaluate the efficacy of guselkumab compared to an inactive drug in participants with low body surface area moderate plaque psoriasis and special site involvement.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have a diagnosis of plaque psoriasis (with or without psoriatic arthritis) for at least 6 months before first administration of study intervention
* All participants must meet the following disease severity criteria at screening and at baseline: (a) Overall Investigator's Global Assessment (IGA) 3 (moderate) plaque psoriasis; (b) Body Surface Area (BSA) 2-15 percent (%) with at least 1 plaque outside of special sites; (c) Involvement of at least 1 special site with at least moderate severity. Qualifying sites include scalp with scalp-specific IGA greater than or equal to (>=) 3, face with facial psoriasis IGA >=3, intertriginous with intertriginous psoriasis IGA >=3, or genital with static physician global assessment of genitalia (sPGA-G) >=3
* All participants be inadequately controlled with or intolerant of at least 1 prior topical therapy (including, but not limited to, corticosteroids, retinoids, vitamin D, or vitamin D/steroid and retinoid/steroid combinations, tacrolimus, pimecrolimus, anthralin/dithranol, coal tar preparations, tapinarof, roflumilast, etcetera) for the treatment of psoriasis at both screening
* All participants be a candidate for phototherapy or systemic treatment for psoriasis

Exclusion Criteria:

* Has a nonplaque form of psoriasis (example, erythrodermic, guttate, or pustular) at screening or randomization
* Has current drug-induced psoriasis (for example, a new onset of psoriasis or an exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium)
* For participants with palmoplantar involvement, confounding diagnoses, including, but not limited, to palmoplantar pustulosis, eczematous dermatitis, contact/irritant dermatitis, acquired keratoderma, etcetera, should be confirmed and excluded
* Participants will not be eligible if they have ever received prior biologic (or biosimilars of) for the treatment of psoriasis, psoriatic arthritis (PsA), or any other indications that could impact the assessment of psoriasis. Prior biologics (or biosimilars of) may include, but not limited to, tumor necrosis factor (TNF)-inhibitors (for example: adalimumab, etanercept, infliximab, or certolizumab or biosimilars), interleukin (IL)-17 inhibitors (for example: secukinumab, ixekizumab, brodalumab, or bimekizumab), and IL-12/23 inhibitors (for example: ustekinumab), or IL-23 inhibitor (for example: guselkumab, risankizumab or tildrakizumab)
* Has a history of chronic or recurrent infectious disease, including, but not limited to, chronic renal infection, chronic chest infection (for example, bronchiectasis), recurrent urinary tract infection (recurrent pyelonephritis or chronic non-remitting cystitis), fungal infection (mucocutaneous candidiasis), or open, draining, or infected skin wounds or ulcers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve an Investigator's Global Assessment (IGA) Score of Cleared (0) or Minimal (1) at Week 16 | Week 16
  Percentage of participants who achieve an IGA score of cleared (0) or minimal (1) at Week 16 will be reported. The IGA documents the investigator's assessment of the participant's psoriasis. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).

SECONDARY OUTCOMES:
Change From Baseline in Body Surface Area (BSA) Affected With Psoriasis at Week 16 | Baseline, Week 16
  Change from baseline in BSA affected with psoriasis at Week 16 will be reported. The BSA is a measurement of involved skin over the whole body. The overall BSA affected by psoriasis is estimated based on the participant's handprint (defined as the entire palmar surface of the hand including fingers).
Change From Baseline in Total Psoriasis Area and Severity Index (PASI) Score at Week 16 | Baseline, Week 16
  Change from baseline in PASI score at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for erythema, induration and scaling, which are each rated on a scale of 0 to 4 that is none to maximum severity. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease.
Percentage of Participants who Achieve an Investigator's Global Assessment (IGA) Score of Cleared (0) at Week 16 | Week 16
  Percentage of participants who achieve an IGA score of cleared (0) at Week 16 will be reported. The IGA documents the investigator's assessment of the participant's psoriasis. Overall lesions are graded for induration, erythema, and scaling. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Percentage of Participants who Achieve a PASI 90 Response at Week 16 | Week 16
  Percentage of participants who achieve a PASI 90 response at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for erythema, induration and scaling, which are each rated on a scale of 0 to 4 that is none to maximum severity. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response is defined as greater than or equal to (>=) 90 percent (%) improvement in PASI score from baseline.
Percentage of Participants who Achieve a PASI 100 Response at Week 16 | Week 16
  Percentage of participants who achieve a PASI 100 response at Week 16 will be reported. The PASI is a system used for assessing and grading the severity of psoriatic lesions and their response to therapy. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas is assessed separately for erythema, induration and scaling, which are each rated on a scale of 0 to 4 that is none to maximum severity. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 100 response is defined as 100% improvement in PASI score from baseline.
Percentage of Participants who Achieve a Scalp-Specific Investigator Global Assessment (ss-IGA) Score of Absence of Disease (0) or Very Mild Disease (1) at Week 16 Among Participants With an ss-IGA Score >=3 at Baseline | Week 16
  Percentage of participants who achieve a ss-IGA score of absence of disease (0) or very mild disease (1) at Week 16 among participants with an ss-IGA score >=3 at baseline will be reported. The ss-IGA instrument is used to evaluate the disease severity of scalp psoriasis. Scalp lesions are graded for induration, erythema, and scaling. The participant's scalp psoriasis is assessed as absence of disease (0), very mild disease (1), mild disease (2), moderate disease (3), or severe disease (4).
Percentage of Participants who Achieve a Static Physician's Global Assessment of Genitalia (sPGA-G) Score of Clear (0) or Minimal (1) at Week 16 Among Participants With a sPGA-G Score >=3 at Baseline | Week 16
  Percentage of participants who achieve a sPGA-G score of clear (0) or minimal (1) at Week 16 among participants with a sPGA-G score >=3 at baseline will be reported. The sPGA-G is used to evaluate the disease severity of genital psoriasis. Severity of genital psoriasis is determined by a combination of 3 plaque characteristics: erythema, elevation, and scale. The participant's severity of genital psoriasis is assessed as clear (0), minimal (1), mild (2), moderate (3), severe (4), and very severe (5).
Percentage of Participants who Achieve an Intertriginous IGA (i-IGA) Score of Clear (0) or Minimal (1) at Week 16 Among Participants With an i-IGA Score >=3 at Baseline | Week 16
  Percentage of participants who achieve an i-IGA score of clear (0) or minimal (1) at Week 16 among participants with an i-IGA score >=3 at baseline will be reported. The IGA used for the full body assessment has been adapted with descriptions of disease features that are more consistent with intertriginous psoriasis presentation. The intertriginous areas affected to be scored include the axillary, sub-mammary, abdominal fold, inguinal, and intergluteal cleft/peri-anal region (distinct from genital/perineum involvement). The participant's intertriginous areas affected are assessed as clear (0), minimal (1), mild (2), moderate (3), and severe (4).
Percentage of Participants who Achieve a Facial IGA (f-IGA) Score of Clear (0) or Minimal (1) at Week 16 Among Participants With an f-IGA Score >=3 at Baseline | Week 16
  Percentage of participants who achieve a f-IGA score of clear (0) or minimal (1) at Week 16 among participants with an f-IGA score >=3 at baseline will be reported. The IGA used for the full body assessment will be adapted for use, but only the face will be scored. The participant's facial psoriasis is assessed as clear (0), minimal (1), mild (2), moderate (3), and severe (4).
Change From Baseline in Psoriasis Symptom and Sign Diary (PSSD) Total Symptom Score at Week 16 | Baseline, Week 16
  Change from baseline in PSSD total symptom score at Week 16 will be reported. The PSSD includes patient-reported outcome (PRO) questionnaire designed to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. The PSSD is a patient-reported outcome instrument that includes 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores are derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants who Achieve >=4 Point Reduction (Improvement) in PSSD Itch Score From Baseline at Week 16 Among Participants With a PSSD Itch Score >=4 at Baseline | Week 16
  Percentage of participants who achieve >=4 point reduction (improvement) in PSSD itch score from baseline at Week 16 among participants with a PSSD itch score >=4 at baseline will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit The PSSD is a patient-reported outcome instrument that includes 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores are derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Percentage of Participants With PSSD Individual Symptom Scale Score of 0 at Week 16 Among Participants With PSSD >0 at Baseline | Week 16
  Percentage of participants with PSSD individual symptom score of 0 at Week 16 among participants with PSSD >0 at baseline will be reported. The PSSD includes PRO questionnaire designed to measure the severity of psoriasis symptoms and signs for the assessment of treatment benefit. The PSSD is a patient-reported outcome instrument that includes 11 items covering symptoms (itch, pain, stinging, burning and skin tightness) and participant observable signs (skin dryness, cracking, scaling, shedding or flaking, redness and bleeding) using 0 to 10 numerical rating scales for severity. Two sub scores are derived each ranging from 0 to 100: the psoriasis symptom score and the psoriasis sign score. A higher score indicates more severe disease.
Number of Participants With Adverse Events (AEs) | Up to Week 56
  Number of participants with AEs will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants With Serious Adverse Events (SAEs) | Up to Week 56
  Number of participants with SAEs will be reported. A SAE is any untoward medical occurrence that may results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (64):
- United States (45):
  - Total Dermatology, Birmingham, Alabama
  - Cahaba Research Inc, Birmingham, Alabama
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology, Fountain Valley, California
  - Practice Wang, Riverside, California
  - Therapeutics Clinical Research, San Diego, California
  - Rehlen, Bartlow, Goodman and Baron Dermatology Group, Santa Ana, California
  - Clinical Science Institute, Santa Monica, California
  - University of Conn Health Center, Farmington, Connecticut
  - TrueBlue Clinical Research, Brandon, Florida
  - Florida Academic Dermatology Centers, Coral Gables, Florida
  - Revival Research, Doral, Florida
  - Glick Research Institute, Margate, Florida
  - Miami VA Healthcare System, Miami, Florida
  - Tory P Sullivan M D PA, North Miami Beach, Florida
  - Atlanta Biomedical Clinical Research, Atlanta, Georgia
  - Kindred Hair and Skin Center, Columbia, Maryland
  - DermAssociates, PC, Rockville, Maryland
  - Lawrence J Green MD LLC, Rockville, Maryland
  - Metro Boston Clinical Partners, Brighton, Massachusetts
  - DermCare, LLC, Quincy, Massachusetts
  - Henry Ford Medical Center, West Bloomfield, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Markowitz Medical OptiSkin, New York, New York
  - Accellacare Research of Cary, Cary, North Carolina
  - Darst Dermatology, Charlotte, North Carolina
  - Piedmont Plastic Surgery and Dermatology, Huntersville, North Carolina
  - Bexley dermatology research, Bexley, Ohio
  - Remington Davis Inc, Columbus, Ohio
  - Apex Dermatology Mayfield Heights, Mayfield Heights, Ohio
  - Dermatology and Laser Center of Charleston, Charleston, South Carolina
  - Palmetto Clinical Trial Services, LLC, Fountain Inn, South Carolina
  - Nashville Skin: Comprehensive Dermatology Center, Nashville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - Bellair Dermatology, Bellaire, Texas
  - Modern Research Associates PLLC, Dallas, Texas
  - Bare Dermatology, Dallas, Texas
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Suzanne Bruce and Associates - The Center for Skin Research, Houston, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Acclaim Dermatology, Sugar Land, Texas
  - Frontier Derm Partners CRO, LLC, Mill Creek, Washington
- Canada (19):
  - Beacon Dermatology, Calgary, Alberta
  - Rejuvenation Dermatology Clinic Edmonton Downtown, Edmonton, Alberta
  - Dr. Chih ho Hong Medical, Surrey, British Columbia
  - Enverus Medical, Surrey, British Columbia
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Brunswick Dermatology Center, Fredericton, New Brunswick
  - CCA Medical Research Corporation, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Centre, Barrie, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - Dr Wei Jing Loo Medicine Professional Corporation, London, Ontario
  - North York Research Inc, North York, Ontario
  - JRB Research Inc, Ottawa, Ontario
  - Canadian Dermatology Center, Toronto, Ontario
  - Toronto Research Centre, Toronto, Ontario
  - FACET Dermatology, Toronto, Ontario
  - Research Toronto, Toronto, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - The Centre de recherche Saint-Louis, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency